CLINICAL TRIAL: NCT06575413
Title: Investigating the Role and Electrophysiological Characteristics of the Human Claustrum Based on SEEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liankun_Ren, Professor, Xuanwu Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-125-001
Record Dates: First submitted 2024-08-16; First posted 2024-08-28 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Refractory Epilepsy; Consciousness, Loss of
Keywords: Refractory Epilepsy; Consciousness; Claustrum
MeSH Terms: conditions — Drug Resistant Epilepsy; Unconsciousness | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Direct electrical stimulation of the Claustrum (Experimental): The investigators performed direct electrical stimulation of the claustrum in drug-resistant epilepsy patients underwent SEEG monitoring.The investigators observed the neural activities before, during, and after stimulation and the claustrum-cortical network to figure out the role of claustrum in consciousness and its underlying electrophysiological mechanism.
  Interventions: Other: Direct Electrical Stimulation

INTERVENTIONS:
Other: Direct Electrical Stimulation — The patients underwent SEEG with at least one electrode targeting the claustrum. The investigators used the claustrum as a target for both mapping and CCEP, recording changes in cortical electrical activity.

SUMMARY:
This single-center prospective study aims to investigate the electrophysiological characteristics and functions of the human claustrum by analyzing clinical, imaging, and electrophysiological data from 14~65-year-old patients with drug-resistant epilepsy.

DETAILED DESCRIPTION:
Stereoelectroencephalography (SEEG) is a method for recording electrical activity from deep brain structures using implanted depth electrodes to provide a three-dimensional view of neuronal activity.

Direct Electrical Stimulation (DES) is a neurosurgical technique that involves delivering electrical impulses to specific brain regions through implanted electrodes to map critical functional areas and to study the connectivity of brain regions.

This study aims to investigate the electrophysiological characteristics and functions of the human claustrum by analyzing clinical, imaging, and electrophysiological data from patients aged 14 to 65 implanted intracranial electrodes , with a specific focus on electrodes targeting the claustrum. This research forms part of a broader initiative to explore the functions of cortical and subcortical regions based on SEEG.

ELIGIBILITY:
Inclusion Criteria:

1. The patients were diagnosed with drug-resistant epilepsy.
2. The patients underwent stereoelectroencephalography (SEEG) implantation for pre-surgical evaluation of epilepsy, with at least one electrode target reaching the claustrum
3. Participants/parents/legal guardian provide informed consent for inclusion

Exclusion Criteria:

1. Subjects that experience surgical complications during the implant procedure will be excluded from the study

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-05-27 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Patients Clinical responses Rating | During the trial(up to 3 hours for each subject)
  Researchers categorized patients' clinical responses as normal, mild, moderate, or severe based on their subjective clinical response.
EEG power in spectral frequency bands | During the trial(up to 3 hours for each subject)
  Using SEEG-implanted electrodes, the investigators applied electrical stimulation of varying intensities to the CLA while observing and recording EEG power changes across six spectral frequency bands during the pre-stimulation, stimulation, and post-stimulation periods.
  EEG Frequency Bands
  * delta (1-4 Hz)
  * theta (5-8 Hz)
  * alpha (9-12 Hz)
  * beta (13-30 Hz)
  * low gamma (31-70 Hz)
  * high gamma (71-150 Hz)
The root mean square (RMS) value of Claustrum-Cortical Evoked Potentials | During the trial(up to 3 hours for each subject)
  All cortical-evoked responses were averaged by time-locking the recordings to the onset of each electrical stimulus (zero) off-line, within a time window of -200 to +400 mses, to quantify the morphology.
  The N1 peak, identified as the first negative deflection distinguishable from the stimulus artifact, was the primary focus due to its clear visibility and reproducibility across different stimulations.
  The root mean square (RMS) value will be calculated for different cortical locations during time windows that encompass both the N1 peak(early response time time window) and the baseline.
  A paired one-sample t-test will be used to compare the RMS values in the early response time window across different cortical sites with the RMS values in the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Liankun Ren, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital,Capital Medical University, Beijing, Beijing Municipality, China